CLINICAL TRIAL: NCT03009695
Title: Impact of Deep Transcranial Magnetic Stimulation (dTMS) on Satiety and Weight Control
Brief Title: Transcranial Magnetic Stimulation (TMS) in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Anna Ferrulli, M.D., Ph.D, Sub-Investigator, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMT/obesi
Record Dates: First submitted 2016-12-04; First posted 2017-01-04 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Food Craving; Appetite and General Nutritional Disorders
Keywords: Transcranial Magnetic Stimulation; Obesity; Food Craving; Appetite/Satiety Hormones; fMRI; Intestinal microbiota; Physical activity
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- High frequency repetitive dTMS + Cue (Experimental): 10 obese individuals fulfilling all inclusion/exclusion criteria for the study will be randomized to active high frequency repetitive dTMS treatment with cue.
  Stimulation will be performed 3 times per week, for 5 weeks (15 treatments).
  In this group, stimulation will be performed with the following features:
  Intensity of stimulation: 120% of the resting Motor Threshold (rMT), Frequency: 18 Hz, Duration of the train: 2 sec, Inter-train interval: 20 sec, Trains number: 80, Total pulses: 2880, Total treatment duration: 29.3 min, Cue (sight of food preferred by patient): present.
  Interventions: Device: High frequency repetitive dTMS
- High frequency repetitive dTMS - No Cue (Experimental): 10 obese individuals fulfilling all inclusion/exclusion criteria for the study will be randomized to active high frequency repetitive dTMS treatment without cue.
  Stimulation will be performed 3 times per week, for 5 weeks (15 treatments).
  In this group, stimulation will be performed with the following features:
  Intensity of stimulation: 120% of the resting Motor Threshold (rMT), Frequency: 18 Hz, Duration of the train: 2 sec, Inter-train interval: 20 sec, Trains number: 80, Total pulses: 2880, Total treatment duration: 29.3 min, Cue (sight of food preferred by patient): absent.
  Interventions: Device: High frequency repetitive dTMS
- Low frequency repetitive dTMS+ Cue (Experimental): 10 obese individuals fulfilling all inclusion/exclusion criteria for the study will be randomized to active low frequency repetitive dTMS treatment with cue.
  Stimulation will be performed 3 times per week, for 5 weeks (15 treatments).
  In this group, stimulation will be performed with the following features:
  Intensity of stimulation: 120% of the resting Motor Threshold (rMT) Frequency: 1 Hz Duration of the train: 10 min Inter-train interval: 1 min Trains number: 4 Total pulses: 2400 Total treatment duration: 43 min Cue (sight of food preferred by patient): present
  Interventions: Device: Low frequency repetitive dTMS
- Low frequency repetitive dTMS - No Cue (Experimental): 10 obese individuals fulfilling all inclusion/exclusion criteria for the study will be randomized to active low frequency repetitive dTMS treatment without cue.
  Stimulation will be performed 3 times per week, for 5 weeks (15 treatments).
  In this group, stimulation will be performed with the following features:
  Intensity of stimulation: 120% of the resting Motor Threshold (rMT), Frequency: 1 Hz, Duration of the train: 10 min, Inter-train interval: 1 min, Trains number: 4, Total pulses: 2400, Total treatment duration: 43 min, Cue (sight of food preferred by patient): absent.
  Interventions: Device: Low frequency repetitive dTMS
- Sham (Sham Comparator): 10 obese individuals fulfilling all inclusion/exclusion criteria for the study will be randomized to sham stimulation.
  Stimulation will be performed 3 times per week, for 5 weeks (15 treatments).
  In this group, stimulation will be performed with the following features:
  Intensity of stimulation: 120% of the resting Motor Threshold (rMT), Frequency: 18 Hz (50% of patients) and 1 Hz (50% of patients), Duration of the train: 2 sec or 10 min, Inter-train interval: 20 sec or 1 min, Trains number: 80 or 4, Total pulses: 2880 or 2400, Total treatment duration: 29.3 or 43 min, Cue (sight of food preferred by patient): present.
  Interventions: Device: Sham

INTERVENTIONS:
Device: High frequency repetitive dTMS — Focal rTMS will be performed using a Magstim Rapid2 magnetic stimulator (The Magstim Co. Ltd., U.K.) equipped with an H-shaped coil. The used H-coil version is the H-addiction specifically designed to stimulate the insula and the Pre-Frontal Cortex (PFC). This novel H-coil allows direct stimulation of deeper brain regions, like insula (3 cm vs 1.5 cm from the skull). Before each stimulation the resting Motor Threshold (rMT) should be determined. The rMT will be determined over the left primary motor cortex, afterwards the coil will be moved forward 6 cm anterior the motor spot and aligned symmetrically over the PFC and insula. Repetitive dTMS induces long-lasting changes in neural excitability and dopamine release, specifically high-frequency rTMS (18 Hz) enhances cortical excitability.
  Arms: High frequency repetitive dTMS + Cue; High frequency repetitive dTMS - No Cue
Device: Low frequency repetitive dTMS — Focal rTMS will be performed using a Magstim Rapid2 magnetic stimulator (The Magstim Co. Ltd., U.K.) equipped with an H-shaped coil. The used H-coil version is the H-addiction specifically designed to stimulate the insula and the Pre-Frontal Cortex (PFC). This novel H-coil allows direct stimulation of deeper brain regions, like insula (3 cm vs 1.5 cm from the skull). Before each stimulation the resting Motor Threshold (rMT) should be determined. The rMT will be determined over the left primary motor cortex, afterwards the coil will be moved forward 6 cm anterior the motor spot and aligned symmetrically over the PFC and insula. Repetitive dTMS induces long-lasting changes in neural excitability and dopamine release, specifically low-frequency rTMS (1 Hz) inhibits cortical excitability.
  Arms: Low frequency repetitive dTMS - No Cue; Low frequency repetitive dTMS+ Cue
Device: Sham — Sham stimulation will be performed by an H-sham-coil. The H-sham-coil is designed to mimic the auditory artifacts and the scalp sensation evoked by the real coil, without stimulating the brain itself. As in the other groups, in each patient the rMT will be determined before each repetitive dTMS session. The sham stimulation will be performed either at high frequency (50% of subjects) or at low-frequency (50% of subjects), according to the previously described methodologies. All obese people in this group will be submitted at the sight of food preferred (cue).
  Arms: Sham

SUMMARY:
Obesity is a metabolic disease that has reached epidemic proportions. Insofar no long-term effective drug treatment was developed for obesity. Lyfe style modulation and bariatric surgery are the only interventions with a limited rate of success. Obesity is due to several factors, mainly linked to a neurophysiological mechanism of "food addiction". The use of repetitive deep Transcranial Magnetic Stimulation (dTMS) was proposed to reduce appetite and food craving in obese subjects, leading eventually to a weight reduction. dTMS was already tested successfully in other forms of addiction (smoking, alcohol, cocaine) and the usefulness of dTMS in the treatment of food addiction, and therefore in obesity, was hypothesized. End-points of this research will be: 1) effect on food craving; 2) acute and chronic effects on blood level of hormones acting on the appetite regulation; 3) chronic effects on body weight. The demonstration that a safe, non-invasive and repeatable methodology can treat obesity reducing food craving and modulating appetite/satiety hormones secretion will constitute a cornerstone in translational medicine of metabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 22-65 years
2. If the patient is taking medications, it must take on a stable dose for at least a month
3. Obesity: ≤ 30 BMI ≤ 45
4. Ability to follow verbal or written instructions.

Exclusion Criteria:

1. Axis-I and II psychiatric disorders according to DSM criteria 5 (such as Major Depression, Bipolar Disorder, or Attention Deficit Disorder)
2. IQ score < 85
3. Organic brain disorders: history of stroke, brain major surgery or head trauma
4. Pregnancy or lactation, absence of medically approved contraceptive methods in females of childbearing potential
5. Serious or poorly controlled diseases (hepatic, renal or hearth failure, atrial fibrillation or other heart rhythm disorders)
6. H yperglycemia - Fasting glucose level > 170 mg/dl
7. Urine drug screen positive for amphetamines, barbiturates, cannabinoids, cocaine metabolites, opiates and phencyclidine
8. Positivity to blood alcohol test
9. Metal in any part of the head, except for dental fillings
10. Implanted infusion pumps
11. Intracardiac devices (pacemakers, heart valves ...)
12. History of diseases whose exacerbation could be fatal (e.g. cardiovascular disease, increased intracranial pressure)
13. History of epilepsy or a family history of epilepsy among first-degree relatives
14. Medications associated with lowered seizure threshold (such as antidepressants, anxiolytics…)
15. Treatment with anti-obesity medications or other medications influencing body weight within 3 month prior to Screening Visit
16. Starting a weight loss plan at any time during data collection for the subject
17. Patients affected by galactosemia, priapism and terminal illness
18. Patients on fluid restriction for SIADH or other conditions
19. Contraindications to perform the Magnetic Resonance Imaging (MRI).

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in food craving levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Food craving will be evaluated by the Food Cravings Questionnaire-Trait (FCQ-T), a self-report multidimensional questionnaire composed of 39 items aimed to investigate food addiction and eating disorders. Total FCQ-T score will be used as a general measure of trait craving; individual FCQ-T scores related to the 9 measured craving dimensions could be useful in identifying and differentiating craving profiles between specific populations. Food craving will be also evaluated at follow-up visit 1 (1 month after the end of treatment), follow-up visit 2 (6 months after the end of treatment), and follow-up visit 3 (1 year after the end of treatment).

SECONDARY OUTCOMES:
Changes in body weight induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To evaluate the effectiveness of repetitive dTMS on body weight, the variation rate in kilograms of body weight between baseline and after 5 weeks will be considered. Body weight will be also evaluated at the 3 follow-up visits.
Changes in Fat Mass (FM) rate induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in body composition, specifically in FM percentage (%), will be evaluated by body densitometry at the end of treatment compared to baseline. FM rate will be also evaluated at the follow-up visit 2
Acute and chronic changes in insulin levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: insulin (microU/mL). Insulin will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in glucagon levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: glucagon (pg/mL). Glucagon will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in ghrelin levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: ghrelin (pg/mL). Ghrelin will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in leptin levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: leptin (ng/mL). Leptin will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in Growth Hormone (GH) levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: GH (ng/mL). GH will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in Adreno-Cortico-Tropic Hormone (ACTH) levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: ACTH (pg/mL). ACTH will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in Thyroid-Stimulating Hormone (TSH) levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: TSH (microUI/mL). TSH will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in Prolactin levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: Prolactin (ng/mL). Prolactin will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in Cortisol levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: Cortisol (microg/dL). Cortisol will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Acute and chronic changes in Neuropeptide Y levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  To identify acute and chronic changes induced by repetitive dTMS on the neuro-endocrine pathway involved in the hunger/satiety balance, the following parameter will be considered: Neuropeptide Y (pg/mL). Neuropeptide Y will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, at end of treatment and at the 3 follow-up visits).
Changes in Beta-endorphin levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in neurophysiological mechanisms involved in satiety will be evaluated by dosing the main neurotransmitters involved in the reward system, like Beta-endorphins (ng/mL). Beta-endorphins will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, end of treatment and follow-up visits).
Changes in Epinephrine levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in neurophysiological mechanisms involved in satiety will be evaluated by dosing the main neurotransmitters involved in the reward system, like Epinephrine (pg/mL). Epinephrine will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, end of treatment and follow-up visits).
Changes in Norepinephrine levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in neurophysiological mechanisms involved in satiety will be evaluated by dosing the main neurotransmitters involved in the reward system, like Norepinephrine (pg/mL). Norepinephrine will be evaluated acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, end of treatment and follow-up visits).
Changes in Glucose levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in glucose metabolism will be evaluated by glucose (mg/dL). Glucose will be measured acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, end of treatment and follow-up visits).
Changes in Glycated Hemoglobin levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in glucose metabolism will be evaluated by Glycated Hemoglobin (mmol/mol). Glycated Hemoglobin will be measured chronically (at baseline, end of treatment and follow-up visits).
Changes in Cholesterol levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in lipid metabolism will be evaluated by Cholesterol (mg/dL). Cholesterol will be measured acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, end of treatment and follow-up visits).
Changes in Triglyceride levels induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in lipid metabolism will be evaluated by Triglycerides (mg/dL). Triglycerides will be measured acutely (before and immediately after the first and the last rTMS sessions) and chronically (at baseline, end of treatment and follow-up visits).

OTHER OUTCOMES:
Changes in Resting Energy Expenditure (REE) induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Changes in REE (Kcal/day) will be evaluated by Indirect Calorimetry. Indirect Calorimetry will be performed at baseline, at the end of treatment and at the follow-up visit 2.
Changes in Activity Energy Expenditure (AEE) induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  AEE (Kcal/die) will be evaluated by an accelerometer. Minutes of activity, number of steps, traveled kilometers measurements will be aggregated to define AEE
Changes in cutaneous temperature induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Abdomen and nail bed of both hands temperature (°C) will be detected by infrared thermography
Changes in food cue-induced activation of specific brain areas induced by repetitive dTMS and detected by Magnetic Resonance Imaging (fMRI) from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  Cue-induced activation of specific brain areas will be evaluated by functional Magnetic Resonance Imaging (fMRI)
Assessment of adverse events | Through study completion, an average of 1 year
  During all the study duration, participants will be asked if they are experiencing any adverse event (AE), serious adverse events (SAE) and un-expected serious adverse event (UESAE). All adverse events will be recorded in clinical record. SAE and UESAE will be communicated to Ethical Committee and Oversight Authorities. Number of participants experiencing adverse events will be recorded.
Changes in gut microbiota composition induced by repetitive dTMS from baseline at 5 weeks | Baseline and end of treatment (5 weeks)
  A fecal sample will be collected at baseline and at the end of treatment (5 weeks) and gut microbiota analysis will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- San Donato Hospital, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strafella AP, Paus T, Barrett J, Dagher A. Repetitive transcranial magnetic stimulation of the human prefrontal cortex induces dopamine release in the caudate nucleus. J Neurosci. 2001 Aug 1;21(15):RC157. doi: 10.1523/JNEUROSCI.21-15-j0003.2001. PMID 11459878
- [Background] Pascual-Leone A, Houser CM, Reese K, Shotland LI, Grafman J, Sato S, Valls-Sole J, Brasil-Neto JP, Wassermann EM, Cohen LG, et al. Safety of rapid-rate transcranial magnetic stimulation in normal volunteers. Electroencephalogr Clin Neurophysiol. 1993 Apr;89(2):120-30. doi: 10.1016/0168-5597(93)90094-6. PMID 7683602
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Zangen A, Roth Y, Voller B, Hallett M. Transcranial magnetic stimulation of deep brain regions: evidence for efficacy of the H-coil. Clin Neurophysiol. 2005 Apr;116(4):775-9. doi: 10.1016/j.clinph.2004.11.008. Epub 2004 Dec 16. PMID 15792886
- [Background] Innamorati M, Imperatori C, Balsamo M, Tamburello S, Belvederi Murri M, Contardi A, Tamburello A, Fabbricatore M. Food Cravings Questionnaire-Trait (FCQ-T) discriminates between obese and overweight patients with and without binge eating tendencies: the Italian version of the FCQ-T. J Pers Assess. 2014;96(6):632-9. doi: 10.1080/00223891.2014.909449. Epub 2014 May 2. PMID 24793741
- [Background] Uher R, Yoganathan D, Mogg A, Eranti SV, Treasure J, Campbell IC, McLoughlin DM, Schmidt U. Effect of left prefrontal repetitive transcranial magnetic stimulation on food craving. Biol Psychiatry. 2005 Nov 15;58(10):840-2. doi: 10.1016/j.biopsych.2005.05.043. Epub 2005 Aug 8. PMID 16084855
- [Background] Val-Laillet D, Aarts E, Weber B, Ferrari M, Quaresima V, Stoeckel LE, Alonso-Alonso M, Audette M, Malbert CH, Stice E. Neuroimaging and neuromodulation approaches to study eating behavior and prevent and treat eating disorders and obesity. Neuroimage Clin. 2015 Mar 24;8:1-31. doi: 10.1016/j.nicl.2015.03.016. eCollection 2015. PMID 26110109
- [Background] Dinur-Klein L, Dannon P, Hadar A, Rosenberg O, Roth Y, Kotler M, Zangen A. Smoking cessation induced by deep repetitive transcranial magnetic stimulation of the prefrontal and insular cortices: a prospective, randomized controlled trial. Biol Psychiatry. 2014 Nov 1;76(9):742-9. doi: 10.1016/j.biopsych.2014.05.020. Epub 2014 Jun 5. PMID 25038985
- [Derived] Ferrulli A, Senesi P, Sonaglioni A, Cannavaro D, Massarini S, Macri C, Cipponeri E, DeFronzo RA, Luzi L. Weight Loss With SGLT2 Inhibitors, Semaglutide, and Transcranial Magnetic Stimulation in Type 2 Diabetes and Obesity. Obesity (Silver Spring). 2026 Feb;34(2):317-322. doi: 10.1002/oby.70105. Epub 2025 Dec 26. PMID 41451880
- [Derived] Devoto F, Ferrulli A, Zapparoli L, Massarini S, Banfi G, Paulesu E, Luzi L. Repetitive deep TMS for the reduction of body weight: Bimodal effect on the functional brain connectivity in "diabesity". Nutr Metab Cardiovasc Dis. 2021 Jun 7;31(6):1860-1870. doi: 10.1016/j.numecd.2021.02.015. Epub 2021 Feb 25. PMID 33853721